CLINICAL TRIAL: NCT04973163
Title: A Phase Ia/Ib, Open-label, Multicentre Dose-escalation and Expansion Study to Investigate the Safety, Pharmacokinetics and Preliminary Efficacy of BI 1823911 as a Monotherapy and in Combination With Other Anti-cancer Therapies in Patients With Advanced or Metastatic Solid Tumours Expressing KRAS G12C Mutation
Brief Title: A Study to Test Different Doses of BI 1823911 Alone and Combined With Other Medicines in People With Different Types of Advanced Cancer With KRAS Mutation
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1472-0001; 2021-000460-29 (EudraCT Number)
Record Dates: First submitted 2021-07-14; First posted 2021-07-22 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumors, KRAS Mutation
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Intervention Model Description: The following parts will be included in this trial:
  * First: Monotherapy Arm
  * After confirmation of safety: Combination Therapy Arm
  Each arm consists of three parts (dose escalation (A), dose confirmation (B), and dose expansion (C)).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Monotherapy Arm (Experimental): Each arm consists of three parts (dose escalation (A), dose confirmation (B), and dose expansion (C).
  Interventions: Drug: BI 1823911; Drug: Midazolam
- Combination Therapy Arm (Experimental): Will be started after confirmation of safety in the Monotherapy Arm. Each arm consists of three parts (dose escalation (A), dose confirmation (B), and dose expansion (C).
  Interventions: Drug: BI 1823911; Drug: BI 1701963

INTERVENTIONS:
Drug: BI 1823911 — BI 1823911
Drug: BI 1701963 — BI 1701963
  Arms: Combination Therapy Arm
Drug: Midazolam — Midazolam - only administered in Part B (dose confirmation) of the Monotherapy Arm
  Arms: Monotherapy Arm

SUMMARY:
This study is open to adults with different types of advanced or metastatic cancer (including lung cancer, colorectal cancer, pancreatic cancer, and bile duct cancer). This study is for people for whom previous treatment was not successful or no treatment exists.

People who have a tumour with a KRAS mutation can participate in the study. A KRAS mutation makes tumours grow faster. BI 1823911 and BI 1701963 are medicines that may turn off KRAS, each in a different way. In this study, BI 1823911 is given to people for the first time.

The purpose of this study is to find the highest dose of BI 1823911 that people can tolerate when taken alone and together with BI 1701963. The most suitable dose is used to find out whether BI 1823911 alone and in combination with BI 1701963 can make tumours shrink.

Participants can stay in the study as long as they benefit from treatment and can tolerate it.

During this time, participants take tablets of BI 1823911 alone or in combination with BI 1701963 once a day. The doctors regularly monitor the size of the tumour. Doctors also regularly record any unwanted effects and check participant's health.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of locally advanced or metastatic solid tumours, e.g. adenocarcinoma of the lung, colorectal cancer, pancreatic cancer or cholangiocarcinoma. Non-small cell lung cancer (NSCLC) patients with mixed histology are eligible if adenocarcinoma is the predominant histology.
* Documented disease progression despite appropriate prior standard therapies or for whom no standard therapy exists for their tumour type and disease stage.
* KRAS mutation status: Kirsten rat sarcoma virus homolog (KRAS) glycine-to-cysteine (G12C) mutation in tumour tissue or blood based on previously performed local testing using a validated test.
* Provision of archival tumour tissue, if available, to confirm retrospectively KRAS G12C mutation status and for biomarker assessment.
* At least one target lesion that can be measured per Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1 (radiated lesions do not qualify as target lesions). In patients who only have one target lesion, and a biopsy of the lesion is required, the baseline imaging must be performed before the biopsy or at the earliest two weeks after the biopsy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ function as follows:

  * Absolute neutrophil count (ANC) ≥1.5 x 10^9/L (equivalent values: ≥ 1.5 x 10³/μL or ≥ 1500/mm³); hemoglobin ≥9.0 g/dL (equivalent values: ≥ 90 g/L or ≥ 5.6 mmol/L); platelets ≥100 x 10^9/L (equivalent values: ≥ 100 x 10³/μL or ≥ 100 x 10³/mm³) without the use of haematopoietic growth factors.
  * Total bilirubin ≤1.5 times the upper limit of normal (ULN), or ≤4 x ULN for patients who are known to have Gilbert's syndrome.
  * Creatinine ≤1.5 x ULN. If creatinine is >1.5 x ULN, patient is eligible if concurrent creatinine clearance ≥50 mL/min (equivalent value: 0.84mL/s) (measured or calculated by Cockcroft-Gault formula).
  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤3 x ULN, for patients with liver metastases ≤5 x ULN.
* Age ≥18 years of age, or over the legal age of consent as required by local legislation.

Further inclusion criteria apply.

Exclusion Criteria:

* Previous anticancer chemotherapy within 3 weeks of the first administration of trial drug. Previous anticancer hormonal treatment or anticancer immunotherapy within 2 weeks of the first administration of trial drug.
* Previous treatment with Rat Sarcoma (RAS), Mitogen-activated protein kinase (MAPK) or Son of sevenless 1 (SOS1) targeting agents (only for monotherapy Parts A, B, and C).
* Radiotherapy within 2 weeks prior to start of treatment, provided recovery from related toxicity.
* Major surgery (major according to the investigator's assessment) performed within 4 weeks prior to start of treatment or planned during the projected course of the trial, e.g. hip replacement.
* Previous treatment with any investigational agent(s) or targeted treatment within 28 days prior to start of treatment or 5 half-lives, whichever is shorter.
* Known history of hypersensitivity to any of the excipients of BI 1823911 tablets, or any contraindication to Midazolam (for Monotherapy Part B only).
* History or presence of cardiovascular abnormalities such as congestive heart failure New York Heart Association (NYHA) classification of ≥3, unstable angina or poorly controlled arrhythmia which are considered clinically relevant by the Investigator. Myocardial infarction within 6 months prior to start of treatment. Uncontrolled hypertension defined as: Blood pressure (BP) measured in a rested and relaxed condition, where systolic BP >=140 mmHg, or diastolic BP >= 90 mmHg, with or without medication.
* Left ventricular ejection fraction (LVEF) <50%. Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2026-11-29 (Estimated); Study Completion 2026-12-27 (Estimated)

PRIMARY OUTCOMES:
Dose escalation (Part A) - Monotherapy and combination therapy: Number of patients experiencing Dose limiting toxicities (DLTs) during the Maximum tolerated dose (MTD) evaluation period for BI 1823911 in monotherapy and in each combination | up to 28 days
  DLTs are graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Dose confirmation (Part B) and expansion (Part C) - Monotherapy and combination therapy: Objective response (OR) defined as best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR) | up to 39 months
  BOR is determined according to Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1.
  BOR will consider all tumour assessments from first treatment administration until the earliest of disease progression, death, or last evaluable tumour assessment before start of subsequent anti-cancer therapy, loss to follow-up, or withdrawal of consent.

SECONDARY OUTCOMES:
Dose escalation (Part A) - Monotherapy and combination therapy: Number of patients experiencing DLTs during all treatment cycles for BI 1823911 in monotherapy and in each combination | up to 39 months
Dose confirmation (Part B) and expansion (Part C) - Monotherapy and combination therapy: Objective response (OR) | up to 39 months
  OR is defined as best overall response (BOR) of complete response (CR) or partial response (PR), both regardless of confirmation.
  BOR is determined according to RECIST version 1.1. BOR will consider all tumour assessments from first treatment administration until the earliest of disease progression, death, or last evaluable tumour assessment before start of subsequent anti-cancer therapy, loss to follow-up, or withdrawal of consent.
Dose confirmation (Part B) and expansion (Part C) - Monotherapy and combination therapy: Duration of OR | up to 39 months
  Duration of OR is defined as the time from first documented CR or PR until disease progression or death (whichever occurs first) among patients with OR.
Dose confirmation (Part B) and expansion (Part C) - Monotherapy and combination therapy: Tumour shrinkage (in millimetres) | up to 39 months
  Tumour shrinkage is defined as the difference between the minimum post-baseline sum of diameters of target lesions (longest for non-nodal lesions, short axis for nodal lesions) and the baseline sum of longest diameters of the same set of target lesions.
Dose confirmation (Part B) and expansion (Part C) - Monotherapy and combination therapy: Progression-free survival (PFS) rate | at month 6
  PFS is defined as the time from first treatment administration until tumour progression according to RECIST version 1.1 or death from any cause, whichever occurs earlier.
All study parts: Number of patients with adverse events during the on-treatment period | up to 39 months
All study parts, BI 1823911: Maximum concentration (Cmax) | up to 24 hours
All study parts, BI 1823911: Steady state concentration (Css) | up to 24 hours
All study parts, BI 1823911: Area under the plasma concentration-time curve from time zero to time t (AUCτ) | up to 24 hours
All study parts, BI 1823911: Area under the plasma concentration-time curve at steady state (AUCss) | up to 24 hours
All study parts, BI 1701963: Maximum concentration (Cmax) | up to 24 hours
All study parts, BI 1701963: Steady state concentration (Css) | up to 24 hours
All study parts, BI 1701963: Area under the plasma concentration-time curve from time zero to time t (AUCτ) | up to 24 hours
All study parts, BI 1701963: Area under the plasma concentration-time curve at steady state (AUCss) | up to 24 hours

CONTACTS AND LOCATIONS:
Locations (9):
- United States (3):
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute at Mary Crowley, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Belgium (4):
  - Brussels - HOSP Jules Bordet, Anderlecht/Brussels-Capital
  - Edegem - UNIV UZ Antwerpen, Edegem/Antwerpen
  - Universitair Ziekenhuis Gent, Gent/Oost-Vlaanderen
  - UZ Leuven, Leuven/Vlaams-Brabant
- Hospital Universitari Vall D Hebron, Barcelona, Spain
- The Christie, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com